CLINICAL TRIAL: NCT02365025
Title: The Effects of a Parental Intervention on Electronic Media Exposure and Sleep Patterns in Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Dept B, HaEmek Medical Center, Israel
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 0075-10-EMC
Record Dates: First submitted 2015-01-25; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Sleep
Keywords: Sleep patterns; Electronic Media Exposure; Parental Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Step 1: Patients and parents enrolment. Step 2: The parents of the children assigned to the experimental group will fill a questionaire related to familial and social background, electronic media exposure and sleep characteristics of their children.
  Step 3: Parents of the children assigned to this group will participate in 6 meetings guides by experts in sleeping disorders. In those meeting the parents will be exposed to sleep disturbances, the importance of sleep habits and the influence of electronic media on sleep and learning.
  Step 4: Re evaluation by questioners after the 6 meetings participation. Step 5: 3 months follow up after the intervention (Meetings).
  Interventions: Other: Meetings guides by experts in sleeping disorders.
- Control group (No Intervention): Step 1: Patients and parents enrolment. Step 2: The parents of the children assigned to the control group will fill a questionaire related to familial and social background, electronic media exposure and sleep characteristics of their children.
  Step 3: Parents of the children assigned to this group will not participate in the meetings as described in the experimental group.
  Step 4: Re evaluation by questioners after the time that the experimental group participated in the meetings.
  Step 5: 3 months follow up.

INTERVENTIONS:
Other: Meetings guides by experts in sleeping disorders. — meetings guides by experts in sleeping disorders. In those meeting the parents will be exposed to sleep disturbances, the importance of sleep habits and the influence of electronic media on sleep and learning.
  Arms: Experimental group

SUMMARY:
Amongst adolescents, there is a gap that widens with age between recommended sleep duration and actual sleep time. Due to this gap, bodily and mental functions such as those related to the metabolic and immune systems, performance, memory, school achievement and creative ability can be harmed. Moreover, lack of sleep involves an increased risk of accidents and injuries, behavior problems and reduced quality of life.

Biological factors that explain changes in sleep patterns include delays in the circadian timing system and in the homeostatic system that regulate sleep and wakefulness. These changes cause a growing and continuous delay in sleep phase during adolescence. In addition, a number of environmental factors affect sleep patterns: variables such as early school start time, increased homework assignments, after-school activities, lack of parental demand for adequate sleep hours, and increased "screen time," or use of electronic media, including television, computer games, internet and cellular phones.

Based on the Parental Style model, the authoritative parenting style is characterized by parents setting high demands on their children on the one hand and displaying high levels of responsiveness to their children on the other. The authoritarian parenting style is characterized by parents setting high demands on their children on the one hand yet displaying low levels of responsiveness to their children on the other. The permissive parenting style is characterized by parents setting low demands on their children and displaying high levels of responsiveness to their children. In several investigations, the authoritative parenting style has been shown to have a positive influence on child development, academic achievement and psychosocial competency, and promoted healthy behaviors in adolescents, such as good eating habits, increased physical activity and a decrease in risky behaviors such as smoking, alcohol abuse, extreme diets and early sexual behavior.

The Conceptual Model views parents as the sole agents of change in their children's life, and focuses on the power of personal example, environmental changes and promotion of the authoritative parental style. The main aim of this research is to evaluate the effectiveness of an intervention program that deals with increasing parents' awareness of the changes that characterize adolescents and encourages the authoritative parental style based on the Parenting Style Model.

DETAILED DESCRIPTION:
Amongst adolescents, there is a gap that widens with age between recommended sleep duration and actual sleep time. Due to this gap, bodily and mental functions such as those related to the metabolic and immune systems, performance, memory, school achievement and creative ability can be harmed. Moreover, lack of sleep involves an increased risk of accidents and injuries, behavior problems and reduced quality of life.

Biological factors that explain changes in sleep patterns include delays in the circadian timing system and in the homeostatic system that regulate sleep and wakefulness. These changes cause a growing and continuous delay in sleep phase during adolescence. In addition, a number of environmental factors affect sleep patterns: variables such as early school start time, increased homework assignments, after-school activities, lack of parental demand for adequate sleep hours, and increased "screen time," or use of electronic media, including television, computer games, internet and cellular phones.

Based on the Parental Style model, the authoritative parenting style is characterized by parents setting high demands on their children on the one hand and displaying high levels of responsiveness to their children on the other. The authoritarian parenting style is characterized by parents setting high demands on their children on the one hand yet displaying low levels of responsiveness to their children on the other. The permissive parenting style is characterized by parents setting low demands on their children and displaying high levels of responsiveness to their children. In several investigations, the authoritative parenting style has been shown to have a positive influence on child development, academic achievement and psychosocial competency, and promoted healthy behaviors in adolescents, such as good eating habits, increased physical activity and a decrease in risky behaviors such as smoking, alcohol abuse, extreme diets and early sexual behavior.

The Conceptual Model views parents as the sole agents of change in their children's life, and focuses on the power of personal example, environmental changes and promotion of the authoritative parental style. This model has been found to be effective in the field of eating disorders but has never been implemented in the field of sleep.

The main aim of this research is to evaluate the effectiveness of an intervention program that deals with increasing parents' awareness of the changes that characterize adolescents and encourages the authoritative parental style based on the Parenting Style Model; it also encourages parents to make environmental changes at home based on the Conceptual Model in order to promote healthy behaviors including healthy sleep patterns and controlled exposure to electronic media in young normative adolescents (ages 10-12) .

Research Hypotheses:

Hypothesis 1: There is a link between availability and the amount of time spent using electronic media. Adolescents who have media devices in their rooms are exposed for longer hours to electronic media compared to those who do not have media devices in their rooms. In addition, there is a link between the availability of the media devices and sleep patterns. Adolescents who have media devices in their rooms will show delayed sleep patterns and shorter sleep durations compared to those who do not.

Hypothesis 2: There is a connection between parental style, sleep patterns and media exposure habits in young adolescents. Children of parents with an authoritative style would exhibit proper sleep patterns and exposure to electronic media; and children whose parents have an authoritarian parental style would have longer sleep durations and less exposure to electronic media compared with other parenting styles. It was assumed that children whose parents exhibit the permissive parental style would have shorter sleep duration and more exposure to electronic media compared to other parenting styles.

Hypothesis 3: There is a connection between sleep patterns, media exposure habits and quality of life in young adolescents. The study will find that better sleep patterns and lower exposure to electronic media are related to higher quality of life in young adolescents.

Hypothesis 4: The intervention program based on the Conceptual Model will lead to an increase in parents' knowledge about the changes that characterize adolescents and will promote the authoritative parental style.

Hypothesis 5: The intervention program will lead to an improvement in healthy behaviors, including better sleep patterns, controlled use of electronic media, better quality of life of young adolescents.

Method The sample included 70 dyads of parents (mostly mothers) and adolescents from schools in the Jezreel Valley. The experimental group and the control group each consisted of 35 participants (35 girls) of average age 10.7 (0.9) years. There were three sessions of data collection: 1. baseline, 2. immediately following intervention, 3. three months post-intervention. Parents and adolescents reported on electronic media consumption, sleep patterns and quality of life. In addition, parents reported on their parenting styles and adolescents wore an ActiGraph (for monitoring their sleep patterns) and filled in a sleep diary for five days. Parents in the experimental group participated in six workshops, while parents in the control group received information regarding healthy sleep habits and the effects of excessive media exposure by mail and were expected to read it on their own.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers aged 10 to 12 years, Hebrew speaking and healthy.
* Hebrew speaking parents.

Exclusion Criteria:

* Teenagers suffering from chronic diseases of diseases that leads to learning disabilities.
* Teenagers who live in homes without exposure to electronical media.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Sleep Habits | Two years
  Sleep Habits measured by: Bedtime hour, sleep latency, wake-up time, total sleep, daytime sleepiness, depressed mood, sleep problem behaviors and morningness-eveningness duration both on weekdays and weekends.

SECONDARY OUTCOMES:
Parents Knowledge regarding Sleep and Media | Two Years
  Parents Knowledge regarding Sleep and Media regarding the importance of sleep in adolescence and issues regarding good sleep hygiene.
Quantity of media exposure | Two years
  Quantity of media exposure including whether or not teenagers have television/computer in their bedroom and the use of television, computer games, internet and total media in hours per day

OTHER OUTCOMES:
Quality of life | Two Years
  Quality of life including physical, emotional, social, psycho-social, school function
Parental Authority | Two Years
  Parental Authority: authoritative, Authoritarian and Permissive parenting style.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — HaEmek Medical Center - Afula - IsRAEL